CLINICAL TRIAL: NCT04988139
Title: Therapeutic Effects of Individualized Educational Training on Preschool Children With Global Developmental Delay
Brief Title: Effects of Educational Training on Children With Developmental Delay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021SKHADR032
Record Dates: First submitted 2021-07-31; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Developmental Delay
Keywords: preschool children; developmental delay; educational training; therapeutic effects
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: A total of 20 children with developmental delays who are receiving traditional rehabilitation programs will be enrolled. The participants will be randomized into two groups, including the intervention group (traditional rehabilitation program with additional educational training) and the control group (traditional rehabilitation program without educational training). The intervention group will receive 1 month of individualized educational training, 50 min per session, 1 session per week, a total of 4 sessions. All of the evaluations will be performed before training, re-evaluated 1 month after completion of treatment, and 3 months after completion of the treatment in the study group. The control group will be evaluated at the baseline, 1 month, and 6 months later, respectively.
Who Masked: Outcomes Assessor
Masking Description: Outcomes measurements will be performed by researchers who are blind to the groups' allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): traditional rehabilitation programs with additional individualized educational training
  Interventions: Other: individualized educational training
- Control group (No Intervention): traditional rehabilitation programs without additional individualized educational training

INTERVENTIONS:
Other: individualized educational training — 50 min per session, one session per week, 4 sessions per month, of individualized educational training to preschool children with developmental delays under traditional rehabilitation programs
  Arms: Intervention group

SUMMARY:
Using a single-blind, randomized controlled design to investigate the additional therapeutic effects of individualized educational training on traditional rehabilitation programs for preschool children with developmental delays.

DETAILED DESCRIPTION:
A total of 20 preschool children with developmental delay who are receiving traditional rehabilitation programs will be enrolled.

The participants will be randomized into two groups, including the intervention group (traditional rehabilitation program with individualized educational training: one time per week, 50 min per session, with a total of 4 sessions in one month) and the control group (traditional rehabilitation program without individualized educational training).

Therapeutic effects, including pediatric daily activity, attention, cognitive function, functional performance, quality of life, and physical functional performance at baseline, after one month of treatment, and 3 months after the treatment, will be evaluated.

The evaluators will be blinded to the group's allocation during the whole course of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* preschool children with a diagnosis of developmental delay, under regular traditional rehabilitation programs, intelligence quotient 70 or greater

Exclusion Criteria:

* age less than 3 or greater than 6 of children diagnosed with developmental delay, under regular traditional rehabilitation programs, intelligence quotient 70 or greater

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of daily activity | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Pediatric Daily Occupation Scale
changes of attention | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Conners Kiddie Continous Performance Test, 2nd edition

SECONDARY OUTCOMES:
change of visual motor integration | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Beery-Buktenica Visual Motor Integration
change of intelligence | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Wechsler Intelligence Scale of children
Changes of functional performance | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Pediatric Outcome Data Collection Instrument
changes of quality of life | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Pediatric Quality of Life Inventory
changes of family impact | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Child Health Questionnaire, parent form 28
changes of walking speed | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  walking speed
changes of chair climbing speed | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  stairs climbing speed
changes of balance | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  one leg standing time
changes of balance and coordination | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  timed up and go test
changes of physical function | score change from baseline to 1 month of treatment, and 3 months after treatment, lower scores mean a worse outcome
  5 times sit to stand test

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No